CLINICAL TRIAL: NCT02580630
Title: Achilles Tendinopathy Treated With Heavy Slow Resistance Training Supplemented With Injection of Glucocorticosteroid or Local Anaesthetic.
Brief Title: Achilles Tendinopathy Treated With Training and Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Finn Elkjær Johannsen, chief physician, MD, specialist in Rheumatology, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-15006579
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Achilles Tendinopathy
Keywords: Strength training, injection, glucocorticoid
MeSH Terms: interventions — Running

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training and glucocorticosteroid (Active Comparator): Patients are instructed to carry out strengthening exercises for the diseased achilles tendon 3 times a week. Physiotherapist will instruct all patients in these heavy slow resistance exercises. First time one week after the first injection, and then every month.
  All patients are informed to a reduction in running and jumping sports for the first 3 months, thereafter slowly progressing to normal sports activity.
  Ultrasound guided injection with glucocorticosteroid: 1ml Lidocain 5 mg/ml and 1 ml methylprednisolone 40mg/ml in Kagers triangle underneath the thickest part of the achilles tendon. Injection is given every months until the tendon pain is markedly diminished (max 3 injections).
  Interventions: Behavioral: Reduction in running and jumping; Other: Training; Drug: Ultrasound guided injection with Glucocorticosteroid
- Training and local anesthetic (Active Comparator): Patients are instructed to carry out strengthening exercises for the diseased achilles tendon 3 times a week. Physiotherapist will instruct all patients in these heavy slow resistance exercises. First time one week after the first injection, and then every month.
  All patients are informed to a reduction in running and jumping sports for the first 3 months, thereafter slowly progressing to normal sports activity.
  Ultrasound guided injection with local anaestethic: 1ml Lidocain 5 mg/ml and 1 ml intralipid (for blinding) in Kagers triangle underneath the thickest part of the achilles tendon. Injection is given every months until the tendon pain is markedly diminished (max 3 injections).
  Interventions: Behavioral: Reduction in running and jumping; Other: Training; Drug: Ultrasound guided injection with local anaestethic

INTERVENTIONS:
Behavioral: Reduction in running and jumping — Advocate to avoid running and jumping sports for the first 3 months, thereafter slowly progressing to normal sport activity.
  Other Names: Impact reduction
Other: Training — Patients are instructed to carry out strengthening exercises for the diseased achilles tendon 3 times a week. Physiotherapist will instruct all patients in these heavy slow resistance exercises. First time one week after the first injection, and then week 3, 6, 10. The patient will register all training on a diary and on an App.
  Other Names: Heavy slow resistance training
Drug: Ultrasound guided injection with Glucocorticosteroid — Ultrasound guided injection in Kagers triangle underneath the thickest part of the achilles tendon with 1ml Lidocain 5 mg/ml and 1 ml methylprednisolone 40mg/ml. Injection is given every months until the tendon pain is markedly reduced (VAS morning pain: 0-20, and VAS training pain: 0-40, and Global recovery rating scale (-5 to +5) is +3 to +5 ). (max 3 injections).
  Other Names: Glucocorticosteroid
  Arms: Training and glucocorticosteroid
Drug: Ultrasound guided injection with local anaestethic — Ultrasound guided injection in Kagers triangle underneath the thickest part of the achilles tendon with 1ml Lidocain 5 mg/ml and 1 ml of intralipid (for blinding). Injection is given every months until the tendon pain is markedly reduced (VAS morning pain: 0-20, and VAS training pain: 0-40, and Global recovery rating scale (-5 to +5) is +3 to +5 ). (max 3 injections).
  Other Names: local anaestethic
  Arms: Training and local anesthetic

SUMMARY:
The purpose of this study is to compare in a randomized double blinded controlled trial the effect of heavy slow resistance exercises combined with ultrasound guided injections with local anesthetic with or without glucocorticosteroid in patients with achilles tendinopathy.

DETAILED DESCRIPTION:
Achilles tendinopathy is a common and often longlasting condition especially in a sports population. The highest incidence is seen in sports involving running and jumping.

As the primary treatment eccentric exercises is recommended and 60-90% will benefit by that. Other studies have shown equal effect of stretching exercises. In a new study heavy slow resistance exercises has proven effective in achilles tendinopathy and the best treatment in lig.patellae tendinopathy.

Injection with glucocorticosteroid is often used in the daily clinic, though inflammation is rarely found. Fredberg 2004 found a good short term effect of glucocorticosteroid injection in an RCT, but no effect in the long term, which the investigators explained by an aggressive rehabilitation with running after a few days. Even though 60-90% will benefit from exercises in efficacy studies, a recent pragmatic effectiveness study by Weetke 2015 found that only 26% did benefit from training alone, but if supplemented by need with 1-3 injections of glucocorticosteroid 76% achieved excellent or good result.

To our knowledge no randomized clinical trials have investigated the combined effect of training and injections. The hypothesis of this study is, that training and slowly progressive rehabilitation combined with glucocorticosteroid injections will have better effect than the same training and rehabilitation combined with injections of local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Midsubstance pain in the achilles tendon
* Symptoms for at least 3 months
* Ultrasound scanning at the first visit shows thickness of the achilles tendon above 7 mm or 20% thicker than the contralateral.
* Patient can read and understand danish

Exclusion Criteria:

* Earlier operations in the foot and leg, that is judged to complicate training
* known arthritis.
* known diabetes
* Leg ulcerations or infections in the foot.
* Judged unable to comply with the training protocol.
* Daily use of pain killers
* Glucocorticosteroid injection to the diseased achilles tendon within the last 6 months.
* Earlier allergic reactions to glucocorticosteroid or local anesthetic.
* Pregnancy or planning to become pregnant
* BMI above 30.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
VISA-A score | 6 month
  VISA-A score is a validated score for patients with achilles tendinopathy. score 0-100.

SECONDARY OUTCOMES:
VISA-A score | 3, 12, 24 months
Global rating scale for recovery | 1, 2, 3, 6, 12, 24 months
  11 point box scale
Ultrasound scanning | 3, 6, 12, 24 months
  measurement of the thickness of the achilles tendon and evaluating the tendon structure and flow on a 4 point scale (Newman grading scale)

OTHER OUTCOMES:
patient pain and exercise diary | week 1,2,3,4,5,6,7,8,9,10,11,12,13
  100 mm VAS score for morning pain (average in the week), 100 mm VAS score for pain during training (average in the week). Compliance to the treatment, Side effects to injections is described.

CONTACTS AND LOCATIONS:
Overall Officials: Finn E Johannsen, MD, Principal Investigator — Institute of Sports Medicine Copenhagen, University of Copenhagen, Denmark; Jens L Olesen, MD, PhD, Principal Investigator — Institute of Sports Medicine Copenhagen, University of Copenhagen, Denmark; Michael S Rathleff, PT, PhD, Study Chair — Research Unit for General Practice in Aalborg, Denmark
Locations (1):
- Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, København NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johannsen F, Olesen JL, Ohlenschlager TF, Lundgaard-Nielsen M, Cullum CK, Jakobsen AS, Rathleff MS, Magnusson PS, Kjaer M. Effect of Ultrasonography-Guided Corticosteroid Injection vs Placebo Added to Exercise Therapy for Achilles Tendinopathy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2219661. doi: 10.1001/jamanetworkopen.2022.19661. PMID 35816306